CLINICAL TRIAL: NCT06964971
Title: Treatment of Transfusion-dependent Nonsevere Aplastic Anemia With Luspatercept: a Multicenter Prospective Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-KLS-046-02
Record Dates: First submitted 2025-05-07; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Transfusion-dependent Non-severe Aplastic Anemia
MeSH Terms: interventions — luspatercept; Deferasirox

STUDY DESIGN:
Intervention Model Description: Control Group: Patients will continue with their original basic treatment regimen for the disease (immunosuppressants, androgens（either alone or in combination）) under observation.
  Treatment Group: In addition to the original basic treatment for the disease, patients will be further divided based on whether iron chelation therapy is used, into two subgroups: Luspatercept monotherapy group and Luspatercept combined with deferasirox group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group1 (Experimental): basic treatment regimen + Luspatercept alone
  Interventions: Drug: Luspatercept
- Treatment Group2 (Experimental): basic treatment regimen + Luspatercept combine with Deferasirox
  Interventions: Drug: Luspatercept combine with Deferasirox

INTERVENTIONS:
Drug: Luspatercept — The recommended starting dose of luspatercept is 1.5 mg/kg administered subcutaneously (SC) once every 3 weeks. Treatment response should be evaluated and dosage adjusted after at least 3 treatment cycles (9 weeks).
  Arms: Treatment Group1
Drug: Luspatercept combine with Deferasirox — The recommended starting dose of luspatercept is 1.5 mg/kg administered subcutaneously (SC) once every 3 weeks. Treatment response should be evaluated and dosage adjusted after at least 3 treatment cycles (9 weeks).
  For patient with platelet counts < 50×10⁹/L:
  Deferasirox dosage: 8-10 mg/kg/day, orally.
  For platelet counts ≥ 50×10⁹/L:
  Deferasirox dosage: 20 mg/kg/day, orally. Discontinue deferasirox if serum ferritin drops below 500 μg/L.
  Arms: Treatment Group2

SUMMARY:
The goal of this clinical trial is to learn whether Luspatercept alone or in combination with Deferasirox can promote hematopoietic function in patients with transfusion-dependent non-severe aplastic anemia, as well as to assess the safety and efficacy of this treatment approach.

The main questions it aims to answer is:

whether the combination therapy of Luspatercept and Deferasirox can improve hemoglobin levels in these patients.

Participants will receive Luspatercept every 3 to 5 weeks based on hemoglobin response, undergo complete blood counts every 1 to 3 weeks, and receive other necessary evaluations as required.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age >= 18 years; 2.According to the "Chinese Guidelines for the Diagnosis and Treatment of Aplastic Anemia (2022 Edition)", the patient must be diagnosed with transfusion-dependent non-severe aplastic anemia (TD-NSAA) and meet the requirement of erythroid hyperplasia in bone marrow aspiration from the posterior iliac crest and/or sternum being more than 15%; 3.If not newly diagnosed with TD-NSAA, and there are combined primary disease maintenance medications, the following conditions must be met:

  1. The patient has not received and does not consider HSCT or ATG treatment for at least the next six months;
  2. If maintaining oral immunosuppressive therapy, the course must be at least 6 months and assessed as ineffective;
  3. If maintaining androgen therapy, the course must be at least 3 months and assessed as ineffective;
  4. If maintaining recombinant human erythropoietin therapy, the course must be at least 3 months and assessed as ineffective;
  5. If maintaining thrombopoietin receptor agonist (TPO-RA) therapy, the duration must be >=6 months with confirmed inefficacy, and a washout period of >=1 month is required before study enrollment;
  6. If the above maintenance medication durations are not met, a washout period of at least 1 month is required; 4.Serum ferritin level >= 1000 ng/ml; 5.Complete whole exome sequencing and MDS/AA next-generation sequencing testing are required.

Exclusion Criteria:

* 1. Severe hepatic dysfunction (ALT or AST ≥ 3 × ULN); 2.Severe renal impairment (eGFR < 30 ml/min/1.73m² or patients with end-stage renal disease); 3.Cardiac disease, including New York Heart Association (NYHA) Class 3 or higher heart failure, or severe arrhythmia requiring treatment, or recent myocardial infarction within 6 months of randomization; 4.Patients with uncontrolled hypertension, with controlled hypertension according to NCI CTCAE version 5.0 considered as ≤ Grade 1 for this protocol; 5.Patients with a PNH clone > 1%; 6.Patients planning to become pregnant or who are pregnant; 7.Surgical or clinical conditions that may significantly alter drug absorption, distribution, metabolism, or excretion (e.g., gastritis, ulcers, history of gastrointestinal or rectal bleeding; history of major gastrointestinal surgery); 8.Patients carrying congenital bone marrow failure-related gene mutations (homozygous or heterozygous, regardless of whether they are pathogenic/benign/likely benign/ of uncertain significance).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | Baseline (1 month before treatment), treatment phase: 12 weeks (twice weekly in weeks 1 / 2, once weekly in week 3, once every 3 weeks ), mid-treatment phase: 12 weeks (once every 3 weeks), follow-up period: 48 weeks (once every 12 weeks).
  Mild anemia: Defined as a hemoglobin level <120 g/L in adult males or <110 g/L in adult females, but >90 g/L.
  Moderate anemia: Hemoglobin level between 60-90 g/L. Severe anemia: Hemoglobin level between 30-60 g/L. Extremely severe anemia: Hemoglobin level <30 g/L.

SECONDARY OUTCOMES:
platelets | Baseline (30 days before treatment), treatment phase: 12 weeks (twice weekly in weeks 1 / 2, once weekly in week 3, once every 3 weeks ), mid-treatment phase: 12 weeks (once every 3 weeks).
Ferritin | Baseline (30 days before treatment), treatment phase: 12 weeks ( once every 3 weeks ), mid-treatment phase: 12 weeks (once every 3 weeks)
Proportion of patients transfusion-free for ≥8 weeks and ≥12 weeks | treatment phase: 12 weeks (twice weekly in weeks 1 / 2, once weekly in week 3, once every 3 weeks ), mid-treatment phase: 12 weeks (once every 3 weeks)
Overall response rate (ORR; CR + PR) at Week 12 and Week 24 of treatment | Week 12 and Week 24
  ORR: Overall Response Rate (defined as the proportion of patients achieving complete response [CR] or partial response [PR]).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No